CLINICAL TRIAL: NCT05902039
Title: MRI Study of Blood-brain Barrier Function in CADASIL
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-715
Record Dates: First submitted 2023-04-21; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Cadasil; Blood Brain Barrier Defect
MeSH Terms: conditions — CADASIL

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CADASIL patients: Inclusion Criteria:
  1. Patients with CADASIL confirmed by gene or/and skin biopsy.
  2. The age range is 20-70 years old.
  3. There is no contraindication to MRI examination, and the informed consent is signed.
  exclusion criteria：
  1. Combined with definite cerebrovascular disease, or combined with brain tumor, brain trauma and other causes of brain diseases.
  2. CADASIL is not confirmed.
  3. There are contraindications to examination or refusal to sign the informed consent.
  Interventions: Other: MRI
- Healthy controls: Inclusion Criteria:
  1. The age range is 20-70 years old.
  2. There is no contraindication to MRI examination, and the informed consent is signed.
  exclusion criteria：
  1. Combined with definite cerebrovascular disease, or combined with brain tumor, brain trauma and other causes of brain diseases.
  2. There are contraindications to examination or refusal to sign the informed consent.

INTERVENTIONS:
Other: MRI — All participants underwent an MR examination on a 3T whole-body Prisma MRI system (Siemens, Erlangen, Germany) with a 64-channel head coil, and a 7T whole-body MAGNETOM MR system (Siemens, Erlangen, Germany) using a 32-channel receive/birdcage transmit head coil (NOVA medical). DP-pCASL, Multi-delay pCASL (MD-pCASL) was acquired to evaluate BBB function and cerebral perfusion. T1-weighted magnetization-prepared rapid gradient echo (T1w-MPRAGE) was scanned at both 3T and 7T for registration in the post-processing workflow. T2-weighted fluid-attenuated inversion recovery (T2w-FLAIR) and T2*-weighted gradient echo (T2*w-GRE) were acquired at 7T for high-resolution structural images and evaluation of lesions.
  Other Names: Cognitive Scale and Clinical Scale Evaluation
  Groups: CADASIL patients

SUMMARY:
Diffusion prepared pseudo-continuous ASL (DP-pCASL) is a newly proposed MRI method to noninvasively measure the function of blood-brain barrier (BBB). The investigators aim to investigate whether the water exchange rate across the BBB, estimated with DP-pCASL, is changed in patients with CADASIL, and to analyze the association between BBB water exchange rate and MRI/clinical features in these patients.

DETAILED DESCRIPTION:
Cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy (CADASIL), caused by NOTCH3 gene mutations, is the most frequent monogenic type of hereditary cerebral small vessel disease (CSVD). The unique pathophysiological mechanisms that small vessel disorders in CADASIL are caused by genetic mutations and that the majority of patients do not combine cerebrovascular disease risk factors make CADASIL an ideal model for studying CSVD, and the imaging findings on CADASIL can be used to diagnose and investigate the etiology of CSVD. While abnormalities in the cerebrovascular structure and hemodynamics have been well demonstrated in CADASIL, the abnormality of the BBB remains controversial. One DCE-MRI study suggested an increase in BBB permeability to gadolinium contrast in CADASIL, whereas no abnormality of BBB was found in subsequent studies in mouse models and patients. The aim of this study was to assess whether BBB function is abnormal in patients with CADASIL using DP-pCASL, which is more sensitive to subtle changes in the BBB compared to DCE-MRI. The investigators hypothesized that the BBB water exchange rate (kw) is reduced in patients with CADASIL compared to controls as assessed by DP-pCASL and that the degree of reduction in BBB water exchange rate correlates with the severity of disease in patients with CADASIL.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CADASIL confirmed by gene or/and skin biopsy.
2. The age range is 20-70 years old.
3. There is no contraindication to MRI examination, and the informed consent is signed.

Exclusion Criteria:

1. Combined with definite cerebrovascular disease, or combined with brain tumor, brain trauma and other causes of brain diseases.
2. CADASIL is not confirmed.
3. There are contraindications to examination or refusal to sign the informed consent.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All CADASIL patients and controls who met the criteria described below and who agreed to participate in this study were enrolled. All CADASIL patients included in this study have been visited at Peking University First Hospital, and the included controls were recruited from the community.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
kw | 30 Minutes
  Post-processing of DP-pCASL data was performed offline using LOFT BBB Toolbox. Head motion was corrected using SPM12 and the temporal fluctuations were minimized by using principal component analysis. DP-pCASL data with the b value of 50 s/mm2 were used to obtain the ASL signal from the tissue and capillary compartments respectively, and kw was quantified by using a single-pass approximation model with total generalized variation regularization.

SECONDARY OUTCOMES:
CBF | 30 Minutes
  Post-processing of MD-pCASL data was performed offline using the BASIL toolkit of FSL. Cerebral blood flow (CBF) were calculated by a custom script using the BASIL toolkit of FSL.
ATT | 30 Minutes
  Post-processing of MD-pCASL data was performed offline using the BASIL toolkit of FSL. Arterial transit time (ATT) were calculated by a custom script using the BASIL toolkit of FSL.
QSM | 30 Minutes
  QSM image reconstruction, including phase pre-processing and estimation of susceptibility maps, followed the default QSMbox (https:// gitlab. com/ acostaj/ QSMbox) pipeline for single-echo, coil-combined data.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] St Lawrence KS, Owen D, Wang DJ. A two-stage approach for measuring vascular water exchange and arterial transit time by diffusion-weighted perfusion MRI. Magn Reson Med. 2012 May;67(5):1275-84. doi: 10.1002/mrm.23104. Epub 2011 Aug 19. PMID 21858870
- [Background] Shao X, Ma SJ, Casey M, D'Orazio L, Ringman JM, Wang DJJ. Mapping water exchange across the blood-brain barrier using 3D diffusion-prepared arterial spin labeled perfusion MRI. Magn Reson Med. 2019 May;81(5):3065-3079. doi: 10.1002/mrm.27632. Epub 2018 Dec 18. PMID 30561821
- [Background] Uchida Y, Kan H, Sakurai K, Arai N, Inui S, Kobayashi S, Kato D, Ueki Y, Matsukawa N. Iron leakage owing to blood-brain barrier disruption in small vessel disease CADASIL. Neurology. 2020 Sep 1;95(9):e1188-e1198. doi: 10.1212/WNL.0000000000010148. Epub 2020 Jun 25. PMID 32586899
- [Background] Walsh J, Tozer DJ, Sari H, Hong YT, Drazyk A, Williams G, Shah NJ, O'Brien JT, Aigbirhio FI, Rosenberg G, Fryer TD, Markus HS. Microglial activation and blood-brain barrier permeability in cerebral small vessel disease. Brain. 2021 Jun 22;144(5):1361-1371. doi: 10.1093/brain/awab003. PMID 34000009
- [Background] Sun C, Wu Y, Ling C, Xie Z, Sun Y, Xie Z, Li Z, Fang X, Kong Q, An J, Wang B, Zhuo Y, Zhang W, Wang Z, Yuan Y, Zhang Z. Reduced blood flow velocity in lenticulostriate arteries of patients with CADASIL assessed by PC-MRA at 7T. J Neurol Neurosurg Psychiatry. 2022 Apr;93(4):451-452. doi: 10.1136/jnnp-2021-326258. Epub 2021 Sep 28. No abstract available. PMID 34583945
- [Background] Li Y, Ying Y, Yao T, Jia X, Liang H, Tang W, Jia X, Song H, Shao X, Wang DJJ, Wang C, Cheng X, Yang Q. Decreased water exchange rate across blood-brain barrier in hereditary cerebral small vessel disease. Brain. 2023 Jul 3;146(7):3079-3087. doi: 10.1093/brain/awac500. PMID 36625892
- [Derived] Li Z, Sun D, Ling C, Bai L, Zhang J, Wu Y, Yuan Y, Wang Z, Wang Z, Zhuo Y, Xue R, Zhang Z. Quantitative modeling of lenticulostriate arteries on 7-T TOF-MRA for cerebral small vessel disease. Eur Radiol Exp. 2024 Nov 5;8(1):126. doi: 10.1186/s41747-024-00512-7. PMID 39499373